CLINICAL TRIAL: NCT05310461
Title: Early Versus Deferred Aortic Valve Replacement in Patients With Moderate Aortic Stenosis Combined With Mitral Regurgitation: a Randomized Clinical Trial
Brief Title: Early Versus Deferred Aortic Valve Replacement in Patients With Moderate Aortic Stenosis and Mitral Regurgitation
Acronym: TIAMAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIAMAR
Record Dates: First submitted 2022-03-25; First posted 2022-04-05 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Aortic Valve Replacement in Patients With Moderate Aortic Stenosis Combined With Mitral Regurgitation
MeSH Terms: interventions — Replantation; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early transcatheter or surgical aortic valve replacement (Experimental): Early transcatheter or surgical aortic valve replacement with or without transcatheter or surgical mitral valve repair/replacement.
  Interventions: Procedure: Transcatheter or surgical aortic valve replacement with or without transcatheter or surgical mitral valve repair/replacement
- Control Intervention (Other): Deferred treatment, with intervention once AVA is ≤1.0 cm2 or if concomitant mitral regurgitation meets an indication for intervention.
  Interventions: Procedure: Deferred treatment, with intervention once AVA is ≤1.0 cm2 or if concomitant mitral regurgitation meets an indication for intervention

INTERVENTIONS:
Procedure: Transcatheter or surgical aortic valve replacement with or without transcatheter or surgical mitral valve repair/replacement — Early transcatheter or surgical aortic valve replacement with or without transcatheter or surgical mitral valve repair/replacement.
  Arms: Early transcatheter or surgical aortic valve replacement
Procedure: Deferred treatment, with intervention once AVA is ≤1.0 cm2 or if concomitant mitral regurgitation meets an indication for intervention — Deferred transcatheter or surgical aortic valve replacement with or without transcatheter or surgical mitral valve repair/replacement.
  Arms: Control Intervention

SUMMARY:
The aim of the present study is to investigate safety and efficacy of early versus deferred aortic valve replacement in patients with moderate aortic stenosis combined with moderate mitral regurgitation.

DETAILED DESCRIPTION:
In more than one-half of all patients with valvular heart disease, more than a single valve is involved. Valvular aortic stenosis coexists with significant mitral valve disease in up to one-third of patients undergoing aortic valve replacement (AVR).

Guidelines for the management of valvular heart disease provide recommendations for isolated valvular lesions; data to guide timing of intervention in patients with multivalvular disease is however scarce. Currently, patients with moderate aortic stenosis (AS) in combination with mitral regurgitation have an indication for aortic valve replacement (AVR) only if the concomitant mitral regurgitation meets an indication for surgery. However, the hemodynamic stress of combined valvular lesions is greater than its individual components, and patients may benefit from early intervention.

Furthermore, the presence of multivalvular heart disease complicates the assessment of individual valvular lesions. In patients with combined AS and mitral regurgitation (MR), increased left ventricular pressure exacerbates the mitral regurgitant volume. Conversely, decreased forward flow across the aortic valve underestimates the severity of aortic stenosis when assessed by a pressure gradient.

Standard cut-off values inadequately reflect the hemodynamic stress in concomitant aortic and mitral valve disease, and recommendations for the timing of valvular replacement fail to account for the complex interplay of multiple valvular lesions.

Timing of intervention in patients with combined AS and MR is therefore challenging and evidence on the optimal timing of intervention is scarce.

Thus, the objective of the present study is to investigate safety and efficacy of early versus deferred aortic valve replacement in patients with moderate aortic stenosis combined with at least moderate mitral regurgitation.

Patients with combined aortic stenosis and mitral regurgitation will be screened for eligibility. If eligible and informed consent is provided, patients will be randomly allocated in a 1:1 ratio to early (within 3 months) or deferred aortic valve replacement (with or without mitral valve intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Moderate native aortic stenosis defined by an aortic valve area (AVA) ≤1.5 cm2 and >1.0 cm2 and transvalvular mean gradient ≥20 mmHg and <40 mmHg.
* Primary or secondary mitral regurgitation (at least moderate) defined by effective regurgitant orifice area (EROA) ≥20 mm2 or regurgitant volume ≥30 ml
* New York Heart Association (NYHA) functional class ≥2

Exclusion Criteria:

* Life expectancy <1 year irrespective of valvular heart disease
* Left ventricular ejection fraction <30% or LVESD >70mm
* Echocardiographic evidence of severe right ventricular dysfunction
* Untreated clinically significant CAD requiring revascularisation
* Moderate or severe aortic regurgitation
* Severe tricuspid valve disease requiring intervention
* Symptomatic patients with severe primary MR who are operable and not high risk
* Patients with severe secondary MR who remain symptomatic despite optimal medical therapy and who are judged appropriate for transcatheter edge-to-edge repair or surgery by the Heart Team
* Transcatheter or surgical treatment of valvular and/or coronary artery disease within 90 days prior to randomization
* COPD with home oxygen therapy
* Estimated or measured systolic PAP >70 mmHg
* Stroke within 30 days prior to the randomization
* Inability to provide written informed consent
* Participation in another cardiovascular trial before reaching the primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be a composite of all-cause death, stroke, and unplanned hospitalization for heart failure related to valvular heart disease at 2 years. | 2 years

SECONDARY OUTCOMES:
All-cause death | 5 years
  Number of all-cause death within study participation
Cardiovascular death | 5 years
  Number of patients with Cardiovascular death within study participation
Neurologic events | 5 years
  Number of patients with stroke, symptomatic hypoxic-ischaemic injury, TIA and evaluation
Hospitalization for heart failure | 5 years
  Number of patients who need hospitalization for heart failure within study participation and evaluation
New-onset atrial fibrillation | 5 years
  Number of patients with new-onset atrial fibrillation within study participation and evaluation
Implantation of a permanent pacemaker | 5 years
  Number of patients with atrioventricular conductance disturbance requiring the implantation of a permanent pacemaker
Aortic or mitral valve re-intervention | 5 years
  Number of patients with Aortic or mitral valve re-intervention within study participation and evaluation
NYHA functional class | 5 years
  Measurement of NYHA functional class within study participation
Days alive out of hospital (DAOH) | 5 years
  Calculation of days alive out of hospital (DAOH) within study participation
The evaluation Health-related quality of life assessment by means of the KCCQ 12 questionnaire | 5 years
  Record the health-related quality of life assessment by means of the KCCQ 12 questionnaire within study participation

OTHER OUTCOMES:
Major vascular complications (VARC-3) | 5 years
  Number of patients with major vascular complications within the study population and evaluation
Cardiac structural complications (major, minor) (VARC-3) | 5 years
  Number of patients with cardiac structural complications within the study population and evaluation
Cerebrovascular events (disabling and non-disabling stroke, and TIA) (VARC-3) | 5 years
  Number of patients with Cerebrovascular events (disabling and non-disabling stroke, and TIA) (VARC-3) within the study population and evaluation
Myocardial infarction | 5 years
  Number of patients with Myocardial infarction within the study population and evaluation
Acute kidney injury (VARC-3) | 5 years
  Number of patients with acute kidney injury (VARC-3) within the study population and evaluation
Access-related non-vascular major complications (VARC-3) | 5 years
  Number of patients with access-related non-vascular major complications (VARC-3) within the study population and evaluation
Bleeding type 3-5 (VARC-3) | 5 years
  Record all bleeding type 3-5 (VARC-3) within the study population
Prosthetic valve endocarditis | 5 years
  Number of patients Prosthetic valve endocarditis within the study population
Prosthetic valve thrombosis | 5 years
  Number of patients prosthetic valve thrombosis within the study population
Valve-related dysfunction requiring reintervention | 5 years
  Number of patients valve-related dysfunction requiring reintervention within the study population

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, Prof. Dr., Principal Investigator — Insel Gruppe AG
Locations (3):
- Switzerland (3):
  - Insel Gruppe AG, Inselspital Bern, Bern
  - University Hospital Geneva (HUG), Geneva
  - Heart Clinic Hirslanden, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah AM, Solomon SD. Valvular heart disease in older adults: seeking an ounce of prevention. Eur Heart J. 2016 Dec 14;37(47):3523-3524. doi: 10.1093/eurheartj/ehw354. Epub 2016 Sep 1. No abstract available. PMID 27590452
- [Background] Khan F, Okuno T, Malebranche D, Lanz J, Praz F, Stortecky S, Windecker S, Pilgrim T. Transcatheter Aortic Valve Replacement in Patients With Multivalvular Heart Disease. JACC Cardiovasc Interv. 2020 Jul 13;13(13):1503-1514. doi: 10.1016/j.jcin.2020.03.052. PMID 32646692
- [Background] Unger P, Pibarot P, Tribouilloy C, Lancellotti P, Maisano F, Iung B, Pierard L; European Society of Cardiology Council on Valvular Heart Disease. Multiple and Mixed Valvular Heart Diseases. Circ Cardiovasc Imaging. 2018 Aug;11(8):e007862. doi: 10.1161/CIRCIMAGING.118.007862. No abstract available. PMID 30354497